CLINICAL TRIAL: NCT05317156
Title: The Effect of Cold Vapor on Intubation-Related Symptoms and Comfort in the Early Postoperative Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Maltepe University (Other)
Responsible Party: Principal Investigator, Dr. Özlem İbrahimoğlu, Assisstant Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IstanbulMU13
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Intubation Complication; Cold; Sore Throat; Cough; Hoarseness; Dysphagia
Keywords: Intubation; Nursing care
MeSH Terms: conditions — Common Cold; Pharyngitis; Cough; Hoarseness; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Patients who were hospitalized for surgical intervention in the supine and prone position and met the sample selection criteria will be included in the experimental and control groups by block randomization method using the random numbers table on the computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prone position-Cold vapor group (Experimental): Cold vapor will be applied to the prone position experimental group patients for 15 minutes in the recovery room. For the study, Nebtime UN600A Ultrasonic Nebulizer Device will be used to apply cold steam to the patients which used in the hospital and calibrated (https://elmaslarmedikal.com.tr/urunler/nebtimeun600aultrasonik-nebulizator/). The parameters to be set on the device for the cold vapor to be applied to the patients in the early postoperative period will be vapor intensity level 5 (1-10), air blowing intensity 5 (1-10), heater intensity 1 (+10C), and timer 15 minutes. The patients will be evaluated by the researchers in terms of sore throat, cough, hoarseness, and dysphagia before and 15 minutes after the cold vapor application in the recovery room and at the 6th, 12th, and 24th hours after the cold vapor application in the postoperative service. In addition, the comfort levels of the patients will be evaluated at the 24th postoperative hour.
  Interventions: Other: Cold vapor
- Supine position-Cold vapor group (Experimental): Cold vapor will be applied to the supine position experimental group patients for 15 minutes in the recovery room. For the study, Nebtime UN600A Ultrasonic Nebulizer Device will be used to apply cold steam to the patients which used in the hospital and calibrated (https://elmaslarmedikal.com.tr/urunler/nebtimeun600aultrasonik-nebulizator/). The parameters to be set on the device for the cold vapor to be applied to the patients in the early postoperative period will be vapor intensity level 5 (1-10), air blowing intensity 5 (1-10), heater intensity 1 (+10C), and timer 15 minutes. The patients will be evaluated by the researchers in terms of sore throat, cough, hoarseness, and dysphagia before and 15 minutes after the cold vapor application in the recovery room and at the 6th, 12th, and 24th hours after the cold vapor application in the postoperative service. In addition, the comfort levels of the patients will be evaluated at the 24th postoperative hour.
  Interventions: Other: Cold vapor
- Prone position-Control group (No Intervention): Patients in the prone position control group will receive standard care that includes all medical and non-medical treatments in the hospital. Nursing care, which is routinely applied to patients in the postoperative period, both in the recovery room and in the service, will be continued within the standard care. The patients will be evaluated by the researchers in terms of sore throat, cough, hoarseness, and dysphagia when they come to the recovery room and at the 6th,12th, and 24th hours after the surgery in the postoperative service. In addition, the comfort levels of the patients will be evaluated at the 24th postoperative hour.
- Supine position-Control Group (No Intervention): Patients in the supine position control group will receive standard care that includes all medical and non-medical treatments in the hospital. Nursing care, which is routinely applied to patients in the postoperative period, both in the recovery room and in the service, will be continued within the standard care. The patients will be evaluated by the researchers in terms of sore throat, cough, hoarseness, and dysphagia when they come to the recovery room and at the 6th,12th, and 24th hours after the surgery in the postoperative service. In addition, the comfort levels of the patients will be evaluated at the 24th postoperative hour.

INTERVENTIONS:
Other: Cold vapor — Before surgery, the socio-demographic data of the patients will be recorded. After surgery, patients will be evaluated in the recovery room for their suitability to participate in the study with the Ramsay sedation scale and the Modified Aldrete Scale. Cold vapor will be applied to the patients for 15 minutes in the recovery room during the postoperative period. The parameters to be set on the device for the cold vapor to be applied to the patients in the early postoperative period will be vapor intensity level 5, air blowing intensity 5, heater intensity 1 (+10C), and timer 15 minutes. The patients will be evaluated by the researchers in terms of sore throat, cough, hoarseness, and dysphagia before and 15 minutes after the cold vapor application in the recovery room and at the 6th,12th, and 24th hours after the cold vapor application in the postoperative service. In addition, the comfort levels of the patients will be evaluated at the 24th postoperative hour.
  Arms: Prone position-Cold vapor group; Supine position-Cold vapor group

SUMMARY:
Endotracheal Intubation (EI) is performed in order to monitor the effectiveness of anesthesia and to control the patient's breathing during the surgery under general anesthesia. In EI, which is an invasive procedure, damage to the larynx and trachea may occur during the placement of the endotracheal tube or due to long-term use. Complications such as postintubation ulcer, laryngeal nerve paresis, arytenoid dislocation may develop in the early period due to EI, and patients may have complaints such as sore throat, swallowing problems, hoarseness, and cough in the postoperative period. This affects the comfort of the patients in the postoperative period. For this reason, it is important to prevent intubation-related symptoms of patients who will undergo surgical intervention before they occur.

DETAILED DESCRIPTION:
Endotracheal Intubation (EI) is performed in order to monitor the effectiveness of anesthesia and to control the patient's breathing during the surgery under general anesthesia. In EI, which is an invasive procedure, damage to the larynx and trachea may occur during the placement of the endotracheal tube or due to long-term use. Complications such as postintubation ulcer, laryngeal nerve paresis, arytenoid dislocation may develop in the early period due to EI, and patients may have complaints such as sore throat, swallowing problems, hoarseness, and cough in the postoperative period. In addition, similar complaints may be encountered after extubation due to the displacement of the cuff of the EI and changes in the cuff pressure during the head and body positioning of the patient for surgical intervention after the EI. In the literature, studies examining the effect of intraoperative patient position on symptoms associated with postoperative intubation are limited. Baran Akkuş and Çaparlar (2020) evaluated the postoperative period of sore throat, hoarseness, dysphagia, and cough by controlling the cuff pressure in patients with hyperextension and supine position, and they did not find a significant difference between the groups. Although the severity of intubation-related complaints, which usually regress within 24 to 72 hours in the postoperative period, varies from patient to patient, it can affect the comfort of the patients in the early postoperative period.

In the literature, there are many studies conducted to relieve the symptoms of sore throat, cough, hoarseness, and dysphagia in patients after extubation. In these studies, pharmacological analgesic agents such as nonsteroidal anti-inflammatory drugs, steroids, opioids, local anesthetics; different anesthetic techniques, the use of different sized endotracheal tubes, intubation after complete muscle relaxation, minimizing cuff pressure, and lubricating gels such as local anesthetics or oral lozenges, sprays and mouthwash solutions are used around or inside the intubation tube cuff. There are many studies in the literature on the successful application of non-pharmacological agents in the treatment of pain. Patients with post-operative throat complaints are recommended to take warm liquids, avoid solid food, suck ice chips, use lozenges, and apply steam. The cold application creates vasoconstriction in the vessels in the area where it is applied, decreases the metabolic rate, and reduces edema. The cold application reduces muscle temperature by reducing the tension sensitivity of muscle spindles with the reflex effect of heat receptors or by inactivating trigger points in the muscles and helps to reduce muscle spasm. Thus, it reduces skin sensitivity by lowering the temperature of nerve fibers and receptors. Cold application is especially beneficial in post-traumatic pain, swelling, and muscle spasm. This affects the comfort of the patients in the postoperative period. For this reason, it is important to prevent intubation-related symptoms of patients who will undergo surgical intervention before they occur. Although it is seen in the literature that pharmacological, non-pharmacological, and herbal methods are applied to reduce postoperative sore throat, cough, hoarseness, and dysphagia, no study has been found examining the effect of the cold steam application on symptoms associated with IE.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Having an ASA score of 1-2
* Not having any respiratory problems before the operation
* Not having a neurological disease related to swallowing
* Not having a sore throat due to cancer and chronic diseases
* Not having hoarseness before surgery
* With endotracheal intubation, the duration of the operation is at least 60 minutes under general anesthesia.
* Having surgery in one of the prone and supine positions
* Getting 2 points from the Ramsay Sedation Scale in the postoperative recovery room.
* Having a Modified Aldrete score of at least 9 in the postoperative recovery room
* To be willing to participate in the study.

Exclusion Criteria:

* To undergo emergency surgery
* Being under the age of 18
* Having an ASA score of 3 and above
* Having any respiratory problems in the preoperative period
* Having a neurological disease related to swallowing
* Having a sore throat due to cancer and chronic diseases
* Having throat surgery
* The duration of the operation is less than 60 minutes
* Having surgery in a position other than the prone and supine positions
* Not agreeing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Cold vapor | First 24 hours after surgery
  The sore throat, one of the intubation-related symptoms of the patients who underwent cold vapor, is decreased compared to those who do not. A score between 0 and 10 is taken from the Visual Analogue Scale (VAS). It is good that the score on the scales has decreased.
Cold vapor | First 24 hours after surgery
  The cough, one of the intubation-related symptoms of the patients who underwent cold vapor, is decreased compared to those who do not. A score between 0 and 4 is taken from the Cough Severity Form (CSF). It is good that the score on the scales has decreased.
Cold vapor | First 24 hours after surgery
  Swallowing, one of the intubation-related symptoms of the patients who underwent cold vapor, is decreased compared to those who do not. A score between 0 and 24 is taken from the Swallowing Impairment Score (SIS). It is good that the score on the scales has decreased.
Cold vapor | First 24 hours after surgery
  The hoarseness, one of the intubation-related symptoms of the patients who underwent cold vapor, is decreased compared to those who do not. A score between 0 and 3 is taken from the Shout's Hoarseness Scale (SHS). It is good that the score on the scales has decreased.
Cold vapor | 24th hour after surgery
  The Perianesthesia Comfort Scale (PCS) of the patients for comfort who underwent cold vapor is decreased compared to those who do not. A score between 24 and 144 is taken from the PCS. It is good that the score from the PCS has increased.

IPD SHARING:
Plan to Share IPD: No
A decision will be made after consultation with other researchers.

REFERENCES:
- [Background] Bulut H, Erden S, Demir SG, Cakar B, Erdogan Z, Demir N, Ay A, Aydin E. The Effect of Cold Vapor Applied for Sore Throat in the Early Postoperative Period. J Perianesth Nurs. 2016 Aug;31(4):291-7. doi: 10.1016/j.jopan.2014.10.005. Epub 2016 Feb 24. PMID 27444760
- [Background] Chang JE, Min SW, Kim CS, Han SH, Kwon YS, Hwang JY. Effect of prophylactic benzydamine hydrochloride on postoperative sore throat and hoarseness after tracheal intubation using a double-lumen endobronchial tube: a randomized controlled trial. Can J Anaesth. 2015 Oct;62(10):1097-103. doi: 10.1007/s12630-015-0432-x. Epub 2015 Jul 7. PMID 26149601
- [Background] Kim D, Jeon B, Son JS, Lee JR, Ko S, Lim H. The changes of endotracheal tube cuff pressure by the position changes from supine to prone and the flexion and extension of head. Korean J Anesthesiol. 2015 Feb;68(1):27-31. doi: 10.4097/kjae.2015.68.1.27. Epub 2015 Jan 28. PMID 25664152
- [Background] Jung TH, Rho JH, Hwang JH, Lee JH, Cha SC, Woo SC. The effect of the humidifier on sore throat and cough after thyroidectomy. Korean J Anesthesiol. 2011 Dec;61(6):470-4. doi: 10.4097/kjae.2011.61.6.470. Epub 2011 Dec 20. PMID 22220223
- [Background] Kim D, Jeong H, Kwon J, Kang S, Han B, Lee EK, Lee SM, Choi JW. The effect of benzydamine hydrochloride on preventing postoperative sore throat after total thyroidectomy: a randomized-controlled trial. Can J Anaesth. 2019 Aug;66(8):934-942. doi: 10.1007/s12630-019-01371-2. Epub 2019 Apr 16. PMID 30993537
- [Background] Komasawa N, Mihara R, Imagawa K, Hattori K, Minami T. Comparison of Pressure Changes by Head and Neck Position between High-Volume Low-Pressure and Taper-Shaped Cuffs: A Randomized Controlled Trial. Biomed Res Int. 2015;2015:386080. doi: 10.1155/2015/386080. Epub 2015 Oct 5. PMID 26509152
- [Background] Paltura C, Guvenc A, Develioglu ON, Yelken K, Kulekci M. Original Research: Aerosolized Lidocaine: Effective for Safer Arousal After Suspension Laryngoscopy. J Voice. 2020 Jan;34(1):130-133. doi: 10.1016/j.jvoice.2018.08.012. Epub 2018 Sep 15. PMID 30227980
- [Background] Stout DM, Bishop MJ, Dwersteg JF, Cullen BF. Correlation of endotracheal tube size with sore throat and hoarseness following general anesthesia. Anesthesiology. 1987 Sep;67(3):419-21. doi: 10.1097/00000542-198709000-00025. No abstract available. PMID 3307536
- [Background] Sahbaz M, Khorshid L. The Effect of Cold Vapor and Ice Cube Absorption in the Early Postoperative Period on Sore Throat and Hoarseness Induced by Intubation. J Perianesth Nurs. 2020 Oct;35(5):518-524. doi: 10.1016/j.jopan.2019.12.007. Epub 2020 May 10. PMID 32402773
- See also: Paltura, C., & Yüceant, G. A. (2018). Kısa süreli endotrakeal entübasyonun ses kalitesi ve aralığına etkisi. Çağdaş Tıp Dergisi, 8(1), 26-28. — https://dergipark.org.tr/en/download/article-file/458973
- See also: Zaman, F., & Karahan, E. (2020). The Effect of Cold Vapor Treated to Thyroidectomy Patients During Early Postoperative Period. Eastern Journal of Medicine, 25(1), 118-125. — https://jag.journalagent.com/ejm/pdfs/EJM-18189-ORIGINAL_ARTICLE-KARAHAN.pdf
- See also: Ghaleb, M. A., Falatah, S., & Al-Amoudi, F. A. (2013). The efficacy of licorice gargle for attenuating postoperative sore throat. Am J Res Commun, 1(11), 379-94. — http://www.usa-journals.com/wp-content/uploads/2013/10/Ghaleb_Vol111.pdf
- See also: AKKUŞ, İ. B., & ÇAPARLAR, C. Ö. (2020). Başın Hiperekstansiyonu Endotrakeal Kaf Basıncını Etkiler mi?. Turkiye Klinikleri J Anest Reanim, 18(1), 1-7. — https://pdfs.semanticscholar.org/6ef9/44253f36d5f11c2b39c42fd0f2b87995c7d7.pdf